CLINICAL TRIAL: NCT06219707
Title: Electro-acupuncture for Irritable Bowel Syndrome With Constipation: a Pilot, Randomized, Double-blinded, Sham-controlled Trial
Brief Title: Electro-acupuncture for Irritable Bowel Syndrome With Constipation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanyang Technological University (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Principal Investigator, Linda Zhong, Assoc Prof, Nanyang Technological University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-2023-451
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Irritable Bowel Syndrome With Constipation
Keywords: Acupuncture; Irritable Bowel Syndrome with Constipation; Microbiota

STUDY DESIGN:
Intervention Model Description: Each patient will be scheduled for a total of 12 treatment sessions, 30 minutes for each session, 2 times a week over 6-week period.
Who Masked: Participant, Outcomes Assessor
Masking Description: After a participant's eligibility is confirmed, a randomization number which corresponds to the group allocation will be provided to the acupuncturist. The clinical assessor and participants will be blinded to the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Electro-Acupuncture group (Experimental): Disposable acupuncture needles (0.30 mm in diameter and 25-40 mm in length) are inserted at a depth of 10-30 mm obliquely into scalp acupuncture points (Baihui, Toulinqi) or straightly into body acupuncture points (Taichong, Zhangmen, Sanyinjiao, Zhongwan, Guanyuan, Tianshu, Zusanli). Electroacupuncture will be applied to the abdominal points at fast and dispersed waves through electric needle stimulator (ES-160 6-Channel Programmable Electro-acupuncture) for 30 min. The intensity is adjusted to a level at which patients feel comfortable. The alternating stimulation is believed to produce maximal biochemical responses in the brain.
  Interventions: Device: Acupuncture needles
- Sham-Acupuncture group (Sham Comparator): Disposable acupuncture needles (0.30 mm in diameter and 25-40 mm in length) are inserted (actual penetration of the skin) at the same way as in the acupuncture group but on sham-acupuncture points (Sham-Baihui, Sham-Toulinqi, Sham-Taichong, Sham-Zhangmen, Sham-Sanyinjiao, Sham-Zhongwan, Sham-Guanyuan, Sham-Tianshu, Sham-Zusanli. The sham points aren't acupuncture points nor located on meridians. Both the electroacupuncture and sham acupuncture groups follow the same procedures, including connection to the stimulator device for the same duration. In the sham group, although no electrical current is delivered, the power switch is turned on and the knobs are manipulated to produce audible clicking sounds, mimicking auditory cues of active treatment.
  Interventions: Device: Acupuncture needles

INTERVENTIONS:
Device: Acupuncture needles — The acupuncture needles and related equipment will have already received approval for routine Traditional Chinese Medicine (TCM) clinical practice in Singapore.

SUMMARY:
The aim of the clinical trial is to evaluate the efficacy and safety of electro-acupuncture for irritable bowel syndrome with constipation (IBS-C) patients. 60 IBS-C patients will be randomized and allocated to either the electro-acupuncture arm or the sham acupuncture arm. We hypothesize that electro-acupuncture would result in superior symptom improvement compared to sham acupuncture. In addition, biological samples (blood, urine, and stool) will be collected during the trial for future exploratory studies. These samples will be used to investigate changes in gut microbiota composition and related metabolites. These analyses aim to explore potential mechanistic links between electro-acupuncture interventions and clinical outcomes in subsequent research. Apart from the IBS-C participants, 30 healthy volunteers aged 21 to 65 years (inclusive) will be recruited to provide blood, urine, and stool samples. These samples will serve as a reference for comparative analyses with those from IBS-C patients before and after electro-acupuncture treatment. The healthy controls will not receive any interventions.

DETAILED DESCRIPTION:
I) Study period:

14 weeks, including 2 weeks of run-in (wash-out), 6 weeks of treatment, and 6 weeks of follow-up. 15 visits will be scheduled for each participant, comprising 2 visits during recruitment and the wash-out period, 12 visits during the treatment period, and 1 visit at the end of the follow-up period.

II) Coding of data:

The trial uses patient-blind technique, which means needles for acupuncture and sham acupuncture will be of identical looking and use same package, conduct blinding according to randomization codes. The study will only be unblinded at final statistical analysis and in final report. In case of emergency code breaking, before code breaking, the investigator should well inform the principal investigator of the corresponding participating site. Investigators who break the codes need to explain the reasons and document on patients' notes. The following circumstances can be considered for an emergency breaking, including, but not limited to: (1) When a SAE happens and is considered to be relevant to experimental medication or placebo; (2) When a serious complication happens.

III) AE/SAE reporting:

All AEs that not meeting the criteria for SAEs will be captured on the case report form (CRF). The details include, but not be limited to: (1) date, (2) event description, (3) time of onset, (4) assessment of severity, (5) relationship to study intervention, and (6) time of resolution/stabilization of the event. All AEs occurring while on study will be documented appropriately regardless of relationship. All AEs will be followed to adequate resolution or stabilization. Any medical condition that is present at the time that the participant is screened will be considered as baseline and not reported as an AE. However, if the study participant's condition deteriorates at any time during the study, it will be recorded as an AE. Changes in the severity of an AE will be documented to allow an assessment of the duration of the event at each level of severity to be performed. AEs characterized as intermittent require documentation of onset and duration of each episode. Regarding SAEs, the study investigator will immediately report to the principal investigator for any SAE. SAEs will be followed until satisfactory resolution or until the investigator deems the event to be chronic or the participant is stable. Other supporting documentation of the event may be requested by the Research Ethics Committee (REC) and should be provided as soon as possible. All SAE must be evaluated by the principal investigator and investigators. Once it happened, principal investigator must submit a SAE report to REC within 24 hours and follow up within 7 days. All AEs and SAEs will be reported to REC in the annual progress report and in the final study report.

IV) Compliance and dropout:

For maximizing participants' compliances, first, the investigators have a thorough consent process for all participants by explaining the details of the study schedule, potential side effects of treatment, the responsibilities the participants needed to take and together with the support and reassurance during the whole study. Second, the investigators have a careful scrutiny (2-week run-in period) to exclude ineligible and low compliance participants before randomization. Third, a special e-mail account and a direct telephone hotline equipping with this clinical trial are ways for the study team to actively communicate with participants and reply enquiries. Moreover, extra-visits will be arranged for participants to see WM doctor or TCM practitioner if participants develop adverse events before the next scheduled visit. If any patient has thoughts of withdrawing or dropping out, he/she will try to determine the reason. The investigators would try to find solution in order to keep the patient in the study.

V) Data collection and management:

Case report forms (CRFs) will be filled in by investigators. Collectable information includes patient identification and demographic data, clinical history, dietary history, personal history, family history, substance use, IBS medical history and clinical examination. Data processing will be conducted in accordance with the following protocol:

1. Verification of CRFs: Investigators need to verify CRFs before inputting.
2. Data verification needs to be conducted successively in the following two steps:

   1. Verify the consistency and logicality of data: Review contents of data range and logicality will be determined by the range of each index and the interrelation. Corresponding software formula will also be applied to assist the data input.
   2. Compare database and CRFs by manual testing. Selectively counter check 10% CRFs with participants' medical notes to check the quality of input and analyze.
3. Data inspection and closure of database: After verifying the validity of established database and statistical protocol, principal investigators will lock the data. The locked data are not allowed to change. Confirmed problems found after locking will be handled in the process of statistical analysis. All mistakes and modification should be recorded and kept properly.

Investigators should keep all trial materials, including acknowledgement of all participants, original informed consent forms with participant's signature, all CRFs and detailed record of medications distribution, which should be provided to ethics committee and drug supervision and administration department for reviewing. All files will be maintained in storage for a period of 7 years after the completion of the clinical trial. Data access during study will be restricted except investigators, ethics committee, and government authority. After the study, all the data will be deidentified and available for sharing upon reasonable request.

VI) Sample size calculation:

The study is the first sham-controlled acupuncture trial that uses the Food and Drug Administration (FDA) recommended end point for IBS-C. The sample size was determined based on the study's purpose, statistical precision, feasibility, and reported improvements in clinical symptoms (abdominal pain, bloating, feeling of incomplete defecation, stool frequency, stool shape) from previous acupuncture studies on IBS-C patients. With an alpha of 0.05, a power of 0.8, a 20% dropout rate, and the potential for missing data, a total sample size of 60 patients (30 in experimental arm and 30 in control arm) is required.

VII) Statistical analysis:

All efficacy and safety analyses will be conducted based on intention-to-treat (ITT) principle. Missing values will be imputed by the last-observation-carried-forward method. The statistical analysis will be performed using the Stata software. The statistical significance will be defined as two-sided P-value of <0.05. Baseline characteristics will be reported as mean (SD). Baseline differences between the groups will be evaluated with the application of Student's t-test for normally distributed continuous variables and non-parametric Mann-Whitney U test for non-normally distributed variables. For categorical variables, chi-squared test or Fisher's exact test will be applied. Comparisons between groups will be conducted by using unpaired t-test for normally distributed data and Mann-Whitney test for non-normally distributed data. Within group differences will be evaluated with paired t-test for normally distributed data and Wilcoxon signed-rank test for non-normally distributed data.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfilment of the Rome IV criteria for IBS-C;
2. Age of 21 to 65 years (inclusive);
3. Weekly average of worst daily abdominal pain score of ≥3 (0-10 scale) for at least 12 weeks before the first visit and during screening period;
4. <3 complete spontaneous bowel movements (CSBMs) per week for at least 12 weeks before the first visit and during screening period;
5. Written informed consent.

Exclusion Criteria:

1. Pregnancy or breast-feeding;
2. Medical history of inflammatory bowel diseases, carbohydrate malabsorption, hormonal disorder, known allergies to food additives, and/or any other serious diseases;
3. History of gastrointestinal tract segment removal or bariatric surgery for obesity;
4. Appendectomy or cholecystectomy within the past 2 months, or other abdominal surgeries within the past 6 months prior to trial enrollment;
5. Unstable medical conditions that could be associated with abdominal pain or discomfort and could potentially influence the assessments in this trial (e.g., chronic kidney disease, endometriosis, lactose intolerance);
6. Diagnosed with primary severe mental illness;
7. Patients who have received acupuncture treatment in last three months, or took concomitant medication with affect gastrointestinal motility or visceral sensation, such as antidiarrheal agent, antidepressant, narcotic analgesic, and anticholinergic;
8. Alcoholism or drug abuse in past 1 year;
9. Having needle phobia or allergy to acupuncture needle materials;
10. Antibiotics and probiotics/prebiotics usage in the previous month;
11. Participating in other clinical studies.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Responders have a decrease in the weekly average of worst abdominal pain scores of ≥30% compared with baseline and a weekly increase of ≥1 CSBM | Baseline (week 2), after treatment period (week 8), end of follow-up (week 14)
  Proportion of patients with a decrease in the weekly average of worst abdominal pain scores of ≥30% and a weekly increase of ≥1 CSBM as compared with the baseline.

SECONDARY OUTCOMES:
Proportion of patients with an improvement of ≥30% in abdominal pain scores | Baseline, week 8, week 14
  Proportion of patients with an improvement of ≥30% in abdominal pain scores from baseline.
Proportion of patients with an average increase of 1 or more spontaneous, complete bowel movements per week | Baseline, week 8, week 14
  Proportion of patients with an average increase of 1 or more spontaneous, complete bowel movements per week as compared with the baseline.
Average number of spontaneous bowel movements, complete spontaneous bowel movements per week | Baseline, week 8, week 14
  Average number of spontaneous bowel movements, complete spontaneous bowel movements per week as compared with the baseline.
Percentage of bowel movements with normal consistency | Baseline, week 8, week 14
  Percentage of bowel movements with normal consistency as compared with the baseline.
Percentage of bowel movements with severe or very severe straining during defecation | Baseline, week 8, week 14
  Percentage of bowel movements with severe or very severe straining during defecation as compared with the baseline.
Median time to the first spontaneous bowel movements, complete spontaneous bowel movements after electro-acupuncture | From first session of electro-acupuncture up to the end of follow-up, approximately 12 weeks
  Median time to the first spontaneous bowel movements, complete spontaneous bowel movements after intake of the first session of electro-acupuncture.
Average number of bisacodyl tablets or enemas used per week | Baseline, week 8, week 14
  Average number of bisacodyl tablets or enemas used per week as compared with the baseline number.
Global assessment of efficacy of treatment with Likert scale | Week 5, week 8, week 14
  Global assessment of efficacy of treatment with Likert scale (range: 1-5) at weeks 5, 8, and 14.
Change from baseline in the IBS-C symtoms using IBS Symptom Severity Scale (IBS-SSS) | Baseline, week 5, week 8, week 14
  IBS-SSS (range: 0-500) is a questionnaire used to assess the severity of symptoms in individuals with Irritable Bowel Syndrome (IBS). It typically includes questions related to abdominal pain, bloating, stool consistency, and the impact of IBS symptoms on daily life. Higher scores on this scale indicate more severe symptoms.
Change from baseline in the IBS-C symtoms using IBS Quality of Life (IBS-QOL) | Baseline, week 5, week 8, week 14
  IBS-QOL (range: 0-100) is a measure designed to assess the impact of IBS on a person's quality of life. It includes questions related to how IBS symptoms affect various aspects of daily functioning, such as physical health, emotional well-being, and social activities. Lower scores on this scale indicate a lower quality of life due to IBS.
Change from baseline in the IBS-C symtoms using Patient Assessment of Constipation Symptoms (PAC-SYM) | Baseline, week 5, week 8, week 14
  PAC-SYM (range for each item: 0-4) is a questionnaire used to evaluate the severity and frequency of constipation-related symptoms in patients. It typically covers symptoms like abdominal discomfort, straining during bowel movements, and incomplete evacuation. Higher scores suggest more severe constipation symptoms.
Change from baseline in the IBS-C symtoms using Constipation Quality of Life (PAC-QOL) | Baseline, week 5, week 8, week 14
  PAC-QOL (range for each item: 0-4) is a measure that assesses the impact of constipation on a person's quality of life. It includes questions about how constipation symptoms affect daily activities, emotional well-being, and overall satisfaction with life. Lower scores indicate a poorer quality of life related to constipation.
Change from baseline in the IBS-C symtoms using Patient Health Questionnaire-15 (PHQ-15) | Baseline, week 5, week 8, week 14
  PHQ-15 (range: 0-30) is a self-report questionnaire that assesses somatic symptom severity in individuals. It includes questions related to various physical symptoms, such as headaches, back pain, and stomach discomfort. It is often used as a screening tool to assess somatic symptom burden, and higher scores indicate a greater presence of somatic symptoms.
Change from baseline in the psychological conditions using Hamilton Depression Scale (HAMD) | Baseline, week 8, week 14
  HAMD (range: 0-52 for HAMD-17) is a clinician-administered questionnaire used to assess the severity of depressive symptoms in individuals with depression. It includes items related to mood, feelings of guilt, sleep disturbances, and physical symptoms. Higher scores indicate more severe depression.
Change from baseline in the psychological conditions using Self-rating Depression Scale (SDS) | Baseline, week 8, week 14
  SDS (range: 20-80) is a self-report questionnaire designed to assess the presence and severity of depressive symptoms from the perspective of the individual. It includes questions about mood, feelings of sadness, and physical symptoms associated with depression. Higher scores suggest greater self-reported depression.
Change from baseline in the psychological conditions using Patient Health Questionnaire (PHQ-9) | Baseline, week 8, week 14
  PHQ-9 (range: 0-27) is a widely used self-report tool for assessing depression. It consists of nine questions that correspond to the criteria for major depressive disorder. Individuals rate the frequency of their symptoms over the past two weeks. Higher scores indicate more severe depression.
Change from baseline in the psychological conditions using General Anxiety Disorder (GAD-7) | Baseline, week 8, week 14
  GAD-7 (range: 0-21) is a self-report questionnaire used to assess the presence and severity of generalized anxiety disorder symptoms. It includes questions related to excessive worry, restlessness, and physical symptoms associated with anxiety. Higher scores indicate greater anxiety.
Change from baseline in the psychological conditions using Hospital Anxiety and Depression Scale (HADS) | Baseline, week 8, week 14
  HADS (range for each subscale: 0-21) is a self-report questionnaire that assesses both anxiety and depression symptoms in individuals, often used in healthcare settings. It includes items related to mood, anxiety, and physical symptoms. It provides separate scores for anxiety and depression.
Change from baseline in the psychological conditions using Visceral Sensitivity Index (VSI) | Baseline, week 8, week 14
  VSI (range: 0-75) is a self-report questionnaire used to assess the degree of visceral hypersensitivity in individuals with conditions like irritable bowel syndrome. It includes questions about gastrointestinal symptoms and discomfort, helping to measure sensitivity to visceral sensations.
Change from baseline in the psychological conditions using Perceived Stress Scale (PSS) | Baseline, week 8, week 14
  PSS (range: 0-40) is a self-report questionnaire that measures an individual's perception of stress in their life. It includes questions about how often one perceives situations as stressful and their ability to cope with stress. Higher scores indicate greater perceived stress.
Patient expectancy and trust in treatment with Likert scale | Week 2, week8, week 14
  Assessment of patient expectancy and trust in treatment with Likert scale (range: 1-5) at weeks 2, 8, and 14. Higher scores suggest greater confidence, satisfaction, trust, and positive perception of the treatment.
Recruitment rate | Baseline
  Number of eligible participants who consent and are enrolled in the study divided by the total number of participants screened for eligibility, reported as a percentage.
Retention rate | Baseline to week 14
  Number of enrolled participants who complete the final study visit divided by the total number of enrolled participants, reported as a percentage.
Adherence to treatment protocols | Baseline to week 14
  Proportion of prescribed treatments completed per participant, calculated as the number of treatment sessions received divided by the number of sessions planned, reported as a percentage.
Completeness and quality of symptom diaries and questionnaire responses | Baseline, week 5, week 8, week 14
  Percentage of symptom diaries and questionnaires that are fully completed with no missing or invalid entries, calculated as the number of complete and valid responses divided by the total number of expected responses.
Number and type of adverse events documented | Baseline to week 14
  Total number and types of adverse events recorded throughout the study, categorized by severity and relatedness to the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Linda LD Zhong, PhD, Principal Investigator — Nanyang Technological University
Locations (1):
- Nanyang Technological University, School of Biological Sciences, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
IPD sharing will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available within 7 years after completion of the clinical trial.
Access Criteria: Individual participant data (IPD) will be made available to qualified researchers upon request. To access the data, researchers must submit a formal request, which will be reviewed and approved by the data sharing committee. Data access will be granted for research purposes only and will require adherence to data use agreements and ethics guidelines.

REFERENCES:
- [Background] Han JS. Acupuncture: neuropeptide release produced by electrical stimulation of different frequencies. Trends Neurosci. 2003 Jan;26(1):17-22. doi: 10.1016/s0166-2236(02)00006-1. No abstract available. PMID 12495858
- [Background] Liu Z, Yan S, Wu J, He L, Li N, Dong G, Fang J, Fu W, Fu L, Sun J, Wang L, Wang S, Yang J, Zhang H, Zhang J, Zhao J, Zhou W, Zhou Z, Ai Y, Zhou K, Liu J, Xu H, Cai Y, Liu B. Acupuncture for Chronic Severe Functional Constipation: A Randomized Trial. Ann Intern Med. 2016 Dec 6;165(11):761-769. doi: 10.7326/M15-3118. Epub 2016 Sep 13. PMID 27618593
- [Background] Camilleri M, Kerstens R, Rykx A, Vandeplassche L. A placebo-controlled trial of prucalopride for severe chronic constipation. N Engl J Med. 2008 May 29;358(22):2344-54. doi: 10.1056/NEJMoa0800670. PMID 18509121
- [Background] Schmulson MJ, Drossman DA. What Is New in Rome IV. J Neurogastroenterol Motil. 2017 Apr 30;23(2):151-163. doi: 10.5056/jnm16214. PMID 28274109
- [Derived] Lam WC, Chen H, Siah KTH, Thakur ER, Zhong LLD. Electro-acupuncture for irritable bowel syndrome with constipation: study protocol of a pilot, randomized, double-blinded, sham-controlled trial. Front Neurol. 2025 Sep 12;16:1632822. doi: 10.3389/fneur.2025.1632822. eCollection 2025. PMID 41018183